CLINICAL TRIAL: NCT00797407
Title: Creatine Supplementation for the Prevention of Statin Myalgia
Brief Title: Effectiveness of Creatine in Preventing Muscle Aching From Cholesterol-Lowering Statin Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: David A. Shewmon MD / Endocrinologist, Cleveland Clinic Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-297
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Hypercholesterolemia; Aches; Cramps; Weakness
Keywords: Hydroxymethylglutaryl-CoA Reductase Inhibitors; Creatine; Adverse Effects; Muscle Toxicity
MeSH Terms: conditions — Hypercholesterolemia; Pain; Muscle Cramp; Asthenia | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Creatine — Creatine 5 gm orally twice a day for 5 days, followed by 5 gm once a day
  Other Names: creatine monohydrate

SUMMARY:
The purpose of this study is to determine of creatine will prevent or treat the muscle toxicity side effect of statin drug therapy, whose symptoms are aching, cramping, and weakness. This is tested in patients who have had this side effect from 3 different statin drugs.

DETAILED DESCRIPTION:
Muscle toxicity is the most common limiting side effect of statin therapy. Biochemical studies have suggested the presence of intramuscular creatine deficiency in patients with muscle toxicity. This is a test of oral creatine supplementation in statin intolerant subjects as a method of preventing the onset of this side effect as well as resolving these symptoms when present during statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* hypercholesterolemia in need of aggressive treatment, defined as a high risk of a vascular event, thus subjects with diabetes, pre-diabetes, or known vascular disease
* intolerance (i.e. muscle toxicity symptoms) of at least 3 statin drugs, each confirmed on rechallenge

Exclusion Criteria:

* history of elevated CPK or rhabdomyolysis while taking a statin,
* CPK levels elevated above the normal range at baseline,
* pregnancy.
* renal insufficiency, defined as a serum creatinine ≥ 2.0 mg/dl.
* history of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Combined visual analog pain scales (0-10) for aching, cramping and weakness | baseline, after 5 days of creatine loading, after 6 weeks of creatine+statin, after up to 6 weeks on statin without creatine, after 4 days of rechallenge with creatine while still on statin

CONTACTS AND LOCATIONS:
Overall Officials: David A Shewmon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Wooster Family Health Center, Cleveland Clinic, Wooster, Ohio, United States